CLINICAL TRIAL: NCT02157922
Title: A Double-blind, Randomized, Placebo-controlled Cross Over Study of Inhaled Alginate Oligosaccharide (OligoG) Administered for 28 Days in Subjects With Cystic Fibrosis
Brief Title: A Phase IIb Study of OligoG in Subjects With Cystic Fibrosis
Acronym: SMR-2984
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AlgiPharma AS (Industry)
Collaborators: Eurostars (Other); Smerud Medical Research International AS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMR-2984
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2016-08

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; mucolytic; mucociliary clearance; lung clearance
MeSH Terms: conditions — Cystic Fibrosis | interventions — oligoG CF-5-20

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alginate oligosaccharide (Active Comparator): Inhalation of a dry powder OligoG in the first treatment period, and of placebo the second period
  Interventions: Drug: alginate oligosaccharide
- Placebo (Placebo Comparator): Inhalation of placebo dry powder in the first treatment period, and OligoG in the second period
  Interventions: Drug: alginate oligosaccharide

INTERVENTIONS:
Drug: alginate oligosaccharide — Inhalation
  Other Names: OligoG

SUMMARY:
The purpose of the study is assessment of efficacy and safety of OligoG as a dry powder formulation, in adult subjects with cystic fibrosis.

DETAILED DESCRIPTION:
The primary objective is to demonstrate efficacy of inhaled OligoG measured by FEV1, and supported by secondary endpoints including Mucociliary Clearance, rheology,microbiology and Quality-of-Life.

The secondary objectives are

1. To demonstrate the safety and tolerability of inhaled OligoG as a dry powder for inhalation after multiple dose administration; and
2. To evaluate patient compliance with treatment.

The design will be randomized, double-blind, placebo-controlled, multi-center, cross-over phase II study. Mucociliary and Cough clearance (MCC) will be an exploratory endpoint in a subset of 24 patients, and Lung Clearance Index (LCI) an exploratory endpoint in another subset of 20 or more patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with a confirmed diagnosis of cystic fibrosis defined by:

  1. Clinical features consistent with the diagnosis of CF AND Sweat chloride ≥60 mmol/L by pilocarpine iontophoresis; OR
  2. Genotypic confirmation of CFTR mutation
* Aged 18 years or older
* Positive microbiological finding of Pseudomonas aeruginosa in expectorated sputum or cough swab within 24 months prior to Screening
* FEV1 between 40%-100%
* At Screening no clinical or laboratory findings suggestive of significant pulmonary illness, other than CF
* Female subjects of child bearing potential and sexually active male subjects must use contraception
* Provision written informed consent

Exclusion Criteria:

* Changes in underlying therapy within the 14 days prior to Day 0. Subjects must be willing to remain on the same underlying stable therapy regimens for the duration of the study until the final follow-up visit.
* Changes in physiotherapy technique or schedule within 14 days prior to Day 0.
* Prohibited medications within 7 days prior to Day 0.
* Pulmonary exacerbation within 28 days of Screening.
* Positive microbiological finding of Burkholderia sp. in expectorated sputum or cough swab documented within 12 months prior to Screening.
* Lactose intolerance/milk allergy.
* On-going acute illness. Subjects must not have needed an outpatient visit, hospitalization or required any change in therapy for other pulmonary disease between Screening and Day 0.
* History of, or planned organ transplantation.
* Treatment for Allergic bronchopulmonary aspergillosis (ABPA).
* Requirement for continuous (24 hour/day) oxygen supplementation.
* Diagnosed with the G551D-mutation, and currently on concomitant treatment with Ivacaftor (Kalydeco).
* Concomitant administration of inhaled mannitol or hypertonic saline within 7 days prior to Day 0 (Visit 2).
* Initiation of cycled, inhaled tobramycin (TOBI) and Colistin less than 4 months prior to Screening (Visit 1). Note: Chronic TOBI and Colistin users are allowed to participate in this study, but subjects who have recently initiated chronic TOBI or Colistin should have at least 2 cycles of TOBI or Colistin respectively in the preceding 4 months before being enrolled in this study. Treatment should be phased in line with the antibiotic treatment.
* Concomitant use of all other marketed antibiotic agents is permitted, providing subjects are willing to remain on the same regimens within the 28 days immediately prior to Day 0 and for the entire duration of the study (until the follow-up visit).
* Clinically significant abnormal findings on haematology or clinical chemistry. In addition, any value ≥ 3 x the upper limit of normal will exclude the subject from participating in the study.
* Subjects unable to perform pulmonary function tests according to the ATS/ERS criteria.
* Pregnant or breast-feeding women. A negative urine pregnancy test must be demonstrated in females of child-bearing potential (Section 4.2.9) at Screening.
* Subjects who have participated in any interventional clinical trial within the 28 days prior to Day 0 (Visit 2).
* Subjects with documented or suspected, clinically significant, alcohol or drug abuse.
* Current malignant disease (with the exception of basal cell carcinoma and cervical neoplasia).
* Any serious or active medical or psychiatric illness, which in the opinion of the Investigator, would interfere with subject treatment, assessment, or compliance with the protocol.
* DPI intolerance, active or placebo

For MCC sites only:

* Smoking. A negative Cotinine test must be demonstrated at Screening
* Subjects who have any non-removable metal objects such as metal plates, screws etc in their head, neck, chest or abdominal area
* Subjects for whom participation in this study will exceed the limits of total radiation exposure allowed in any 12 month period (5 mSv), or will exceed 10 mSv over any three year period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-10; Primary Completion 2017-01 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
FEV1 (Forced Expiratory Volume in 1 second) | 28 days, i.e. start and end of treatment periods
  An improvement in FEV1 during treatment with OligoG as compared to placebo is the primary endpoint of the study.

SECONDARY OUTCOMES:
Mucociliary and cough clearance | 28 days, i.e. start and end of treatment periods
  Mucociliary clearance is assessed by measuring the movement of an inhaled radiotracer up the airways.

OTHER OUTCOMES:
Safety | Screening, day 0, 14, 28, 56, 70, 84 and follow up
  Measurement of vital signs, ECG, blood oxygen saturation and pulmonary function tests. Adverse events and concomitant medications will be recorded, and blood samples will be collected for hematology, clinical chemistry and OligoG concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Tacjana Pressler, PhD MD, Principal Investigator — Rigshospitalet, Denmark
Locations (18):
- Rigshospitalet, Copenhagen, Denmark
- Germany (7):
  - Pediatric Pulmonology and Immunology, Charité Universitätsmedizin, Berlin
  - CF Zentrum Köln, Universitätskrankenhaus Köln, Cologne
  - Medizinische Klinik I, Pneumologie, Uniklinik, Frankfurt
  - Klinik für Pneumologie, CF-Ambulanz, Hanover
  - Mukoviszidose-Zentrum für Erwachsene, Med. Klinik V-Innenstadt (LMU), Münich
  - Pneumologische Praxis Pasing, Münich
  - Center for Pediatric Clinical Studies,, Tübingen
- Oslo University Hospital, Oslo, Norway
- Sweden (2):
  - CF-mottagningen, Sahlgrenska Universitetssjukhuset, Gothenburg
  - Stockholm CF-center, Karolinska Universitetssjukhuset, Stockholm
- United Kingdom (7):
  - Regional Respiratory Centre, Belfast City Hospital, Belfast
  - Papworth Hospital, Cambridge
  - Bio-Images Research Ltd, Basement Medical Block, Within GRI, Glasgow
  - Liverpool Heart and Chest Hospital, Liverpool
  - Royal Brompton and Harefield NHS Foundation Trust, London
  - Queens Medical Centre, Nottingham
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hurley MN, Smith S, Forrester DL, Smyth AR. Antibiotic adjuvant therapy for pulmonary infection in cystic fibrosis. Cochrane Database Syst Rev. 2020 Jul 16;7(7):CD008037. doi: 10.1002/14651858.CD008037.pub4. PMID 32671834